CLINICAL TRIAL: NCT06837571
Title: Assessment of Methadone Dose Taken
Brief Title: Methadone Dose Monitoring With a Remote Medication Monitor
Status: Not yet recruiting | Type: Observational
Sponsor: Cari Health Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: IRB3RMM
Record Dates: First submitted 2025-02-15; First posted 2025-02-20 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Methadone Toxicity; Methadone Overdose; Pain, Chronic; Drug Metabolism, Poor, CYP2D6-Related; Metabolism Medication Toxicity
Keywords: Pharmacokinetics
MeSH Terms: conditions — Chronic Pain; Drug Metabolism, Poor, CYP2D6-Related | interventions — Methadone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — interstitial fluid and fingerstick blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Visit 1: AIM 2 : Determine if an RMM can assess the status of taking a prescribed dose of methadone. To complete this aim, the peak and trough concentrations of a witnessed methadone dose will be assessed in dermal ISF collected through the surface of the skin using existing ISF extraction methods and assessed outside the body via with and dermal ISF dialysis tube and external aptamer switch based fiberoptic sensor continuously for 6 hours. Methadone and protein binding factors are independently assessed in the collected ISF samples using (LC-MS and Lateral Flow Assays). We hypothesize that the methadone peak and trough levels in the blood samples will correlate with the levels of methadone in ISF.
  The Investigators hypothesize that the methadone peak and trough levels in the blood samples will correlate with the levels of methadone in ISF.
  Interventions: Device: ISF Extraction Device 2
- Visit 2: AIM 3: Determine if an RMM can continuously assess the status of taking a prescribed dose of methadone over time. To complete this aim, the pharmacokinetic profile of a witnessed methadone dose will be assessed in ISF dialysate continuously from the surface of the skin using the RMM for up to 12 hours (Aim 3a) and over 3 days (Aim 3b). Methadone will also be assessed over these three time points in the continuously collected ISF samples using LC-MS and Lateral Flow Assays. The Investigators hypothesize that a clinician can recognize a dose taken from the RMM generated measurements of dialyzed ISF.
  Interventions: Diagnostic Test: Measurement of Methadone in the Interstitial Fluid (ISF) before and after prescribed dose taken ex vivo; Drug: Measurement of Methadone in the Interstitial Fluid before and after prescribed dose taken in vivo; Device: ISF Extraction Device 2

INTERVENTIONS:
Diagnostic Test: Measurement of Methadone in the Interstitial Fluid (ISF) before and after prescribed dose taken ex vivo — Measurement of Methadone and its metabolites in interstitial fluid with Liquid Chromatography - Mass Spectroscopy (LC-MS) and Aptamer based Assay
  Other Names: dose taken peak-trough test
  Groups: Visit 2
Drug: Measurement of Methadone in the Interstitial Fluid before and after prescribed dose taken in vivo — Measurement of Methadone and its metabolites in ISF with LC-MS and RMM
  Other Names: In vivo Continuous molecular monitoring
  Groups: Visit 2
Device: ISF Extraction Device 2 — Up to 15 minute periods of continuous ISF collection for analysis
  Other Names: Ascilion

SUMMARY:
Proof of concept: Pilot Study

A Pilot, proof of concept, observational study with a long-term goal to develop a minimally invasive wearable Remote Medication Monitor (RMM) that provides continuous, real-time data on methadone levels in interstitial fluid (ISF). An RMM could be used as a medication adherence monitor and would allow for the physician, counselor, patient, or family member to remotely verify that a physician-prescribed dose has been taken.

DETAILED DESCRIPTION:
The investigator will conduct a non-randomized, non-blinded, feasibility study at a single center in the United States. The study will include up to 20 subjects of an equal number of male and female adults (ages 18-70) who have a prescription for methadone.

In Aim 1, the investigators will determine if an RMM can continuously assess the status of taking a prescribed dose of methadone over time, by inserting the dermal ISF sensing elements into the subjects' abdominal skin. Biosample collections (i.e., ISF, blood) and pharmacokinetic monitoring will occur over a 6-hour period. By completing this aim, the investigator will determine if a physician is able to recognize the pharmacokinetic profile of a taken dose of methadone. The physician will see a dosing curve display generated from dermal ISF dialysis fluid sampling using an external fiberoptic sensor system that is worn continuously on the abdomen similar to continuous glucose monitors.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70
* A prescription for methadone at a dose of 10mg or more for at least one week.
* Taking methadone as prescribed during the last 4 days before consent to participate in the study.

Exclusion Criteria:

* Age <18 or >70
* A condition preventing or complicating ISF collection
* dermatological (skin) condition
* immunodeficiency
* recent blood donation
* anemia
* end stage renal disease
* liver cirrhosis
* cancer
* congestive heart failure
* bleeding diathesis
* tuberculosis (TB)
* Any active severe depression
* suicidal ideation
* mania symptoms
* Pregnancy
* Intending to become pregnant during the course of the study
* Enrolled in a substance use disorder treatment program
* Under a conservatorship.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients taking at least 10mg of methadone per day for chronic pain or opioid use disorder,
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-04-26 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Methadone Concentration in ISF before and after a dose | 1 day
  measure dermal interstitial fluid with LC-MS for methadone before and after a daily dose
Methadone Concentration in blood before and after a dose | 1 day
  measure blood for methadone with LC-MS before and after a daily dose
Concentration of Methadone in ISF with LC-MS versus Fluorescent Aptamer Switch | 2 days
  measure ISF with two procedures (Liquid Chromatography - Mass Spectroscopy and Fluoroscopy
Concentration of Methadone in blood with LC-MS versus Fluorescent Aptamer Switch | 2 days
  measure blood with two procedures (Liquid Chromatography - Mass Spectroscopy and Fluoroscopy
Pearson Correlation of Methadone between ISF and Blood | 2 days
  measure blood and ISF methadone with LC-MS and determine pearson correlation
Pearson Correlation between Fluoroscopy and LC-MS ISF Methadone | 2 days
  measure ISF for methadone by LC-MS and Fluoroscopy and determine Pearson correlation

CONTACTS AND LOCATIONS:
Overall Officials: Charmaine Semenluk, MD, Principal Investigator — Synergy Research Inc.
Locations (1):
- Synergy, Lemon Grove, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Friedel M, Werbovetz B, Drexelius A, Watkins Z, Bali A, Plaxco KW, Heikenfeld J. Continuous molecular monitoring of human dermal interstitial fluid with microneedle-enabled electrochemical aptamer sensors. Lab Chip. 2023 Jul 12;23(14):3289-3299. doi: 10.1039/d3lc00210a. PMID 37395135
- [Background] Gomes NO, Raymundo-Pereira PA. On-Site Therapeutic Drug Monitoring of Paracetamol Analgesic in Non-Invasively Collected Saliva for Personalized Medicine. Small. 2023 Mar;19(12):e2206753. doi: 10.1002/smll.202206753. Epub 2023 Jan 15. PMID 36642790
- [Background] Ribet F, Bendes A, Fredolini C, Dobielewski M, Bottcher M, Beck O, Schwenk JM, Stemme G, Roxhed N. Microneedle Patch for Painless Intradermal Collection of Interstitial Fluid Enabling Multianalyte Measurement of Small Molecules, SARS-CoV-2 Antibodies, and Protein Profiling. Adv Healthc Mater. 2023 May;12(13):e2202564. doi: 10.1002/adhm.202202564. Epub 2023 Feb 21. PMID 36748807
- See also: Cari Health Website — http://www.carihealth.com